CLINICAL TRIAL: NCT07047963
Title: Neuropsychological Evaluation in Intellectual Disability
Brief Title: Neuropsychological Evaluation in Intellectual Disability (ENDI)
Acronym: ENDI
Status: Not yet recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, COQUELET Amelie, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2024- A01565- 42
Record Dates: First submitted 2025-05-22; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Down Syndrome (Trisomy 21); Neuropsychology; Cognitive Aging; Alzheimer Disease; Alzheimer Disease, Early Onset
Keywords: Down Syndrome (Trisomy 21); ENDI; Trisomy 21; neuropsychology; ENDI tests battery
MeSH Terms: conditions — Down Syndrome; Alzheimer Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Trisomy 21 patients: Trisomy 21 patients recruted on Main Phase will perform the ENDI tests in order to assess the acceptability of the subtests (individually) and the full neuropsychological battery
  Interventions: Diagnostic Test: ENDI (Neuropsychological Evaluation in Intellectual Disability)
- Patients with Intellectual Disabilities: Patients with Intellectual Disabilities recruted on Preliminary Phase will be will carry out the ENDI tests in order to evaluate subtest design, ergonomics, understanding of instructions and identify any malfunctions. The observations gathered will enable the principal investigator to refine the digital design of the battery in collaboration with the publishing company.
  Interventions: Diagnostic Test: ENDI (Neuropsychological Evaluation in Intellectual Disability)
- Normotypical volunteers: Normotypical volunteers recruted on Preliminary Phase will be will carry out the ENDI tests in order to evaluate subtest design, ergonomics, understanding of instructions and identify any malfunctions. The observations gathered will enable the principal investigator to refine the digital design of the battery in collaboration with the publishing company.
  Interventions: Diagnostic Test: ENDI (Neuropsychological Evaluation in Intellectual Disability)

INTERVENTIONS:
Diagnostic Test: ENDI (Neuropsychological Evaluation in Intellectual Disability) — This neuropsychological battery comprises 15 subtests designed to assess language, memory, attention and executive skills. By analyzing changes in Trisomy 21 patients performance over time, the neuropsychologist can detect early signs of Alzheimer's disease.
  Other Names: ENDI

SUMMARY:
The goal of this observational study is to evaluate the acceptability ofpatients with trisomy 21 (T21) to perform the full battery of ENDI neurospychological tests and each of the subsets.

In this study, three types of population will be recruted : normotypic volunteers, patients with Intellectual Disability and patients T21carriers.

This study is separated into 2 phases :

* A the preliminary phase : this phase will be used to evaluate subtest design, ergonomics and understanding of instructions, and to identify any malfunctions. The observations gathered will enable the principal investigator to refine the digital design of the battery in collaboration with the publishing company. In this phase, normotypical volunteers and patients with intellectual disabilities will be recruted to perform ENDI test battery.
* A main phase : this phase will enable to answer to the main objective. in this phase, patients with Trisomy 21 aged between 25 and 65 will be recruted to perform ENDI test battery.

DETAILED DESCRIPTION:
Trisomy 21 is a genetic disease resulting from a chromosomal anomaly, due to a triplication, bringing the total number of chromosomes to 47. In addition to physical characteristics, adults with Trisomy 21 (T21) generally have an intelligence quotient (IQ) score suggesting mild (IQ: 50-69) to moderate (IQ: 35-49) intellectual disability (ID), and adaptive functional impairments corresponding to this level of ID severity. Progress in medical and social care has led to a significant increase in life expectancy for trisomy 21 patients. De Graaf, Buckley & Skotko (2021) estimate the number of trisomy 21 patients in France at around 35,000, 42% of whom are aged 40 or over. According to Asselin (2005), by 2030, the number of people with intellectual disabilities (ID) aged over 60 should have doubled.

This raises questions about the ageing of this population, all the more so as it is likely to occur earlier, due to reduced neuronal reserve. For example, signs of aging appear 10 years earlier in people with ID, at around age 55. Moreover, this aging process is said to be accelerated Normal cognitive aging in trisomy 21 patients is poorly characterized in the literature; similarly, there is no consensus regarding prodromal signs of Alzheimer's Disease (AD) in T21. However, the presence of the supernumerary chromosome containing the APP (Amyloid Precursor Protein) gene increases the risk of developing AD: 20% of trisomy 21 patients aged 45 and over develop a major neurocognitive disorder (MNCD), and over 50% by the age of 55. T21 is now considered a genetic form of AD, similar to an autosomal dominant form. Identifying AD in this population is therefore a real challenge, especially as AD is identified as the cause of 70% of deaths in trisomy 21 patients.

In cognitive terms, the precursor signs of AD are impairment of memory and temporo-spatial orientation, followed by impairment of praxis, language and visuo-spatial skills. Other authors suggest an early decline in executive functions. More recently, Startin et al. (2019) show that memory and attention tests are more sensitive in detecting prodromal forms. Establishing a diagnosis of neurodegenerative disease in trisomy 21 patients is important for at least 3 reasons. People with intellectual disabilities are often treated with neuroleptics, whose use is not recommended in AD. It also contributes to the adaptation of medical and social care, as ageing disabled people with AD will experience less frequent difficulties, including behavioural changes. According to the Edinburgh Principles, it is important to "ensure that appropriate diagnostic, assessment and intervention resources and services are available to meet the individual needs and promote the healthy ageing of people with intellectual disabilities and cognitive impairment". Finally, at a time when promising pharmacological treatments for AD are emerging for neurotypical subjects, it seems crucial that trisomy 21 patients, who are more at risk of AD, should be diagnosed as early as possible so that they can ultimately benefit from these new therapies. Neuropsychological assessment plays a crucial role in the diagnostic process, as brain imaging and lumbar puncture for AD biomarkers in cerebrospinal fluid are not always feasible.

However, a number of problems remain:

* Neuropsychological assessment is conditioned by the severity of the intellectual disability and the level of literacy/numeracy.
* Few adapted tests are available in French. Tests used in the general population are not transposable, and those based on child assessment batteries are infantilizing.
* Few tests incorporate the evolution of digital technologies, which make it possible to offer more playful interfaces with better temporal control.
* Few tests allow for longitudinal follow-up (no parallel versions, no longitudinal standards), whereas current recommendations call for systematic annual follow-up from the age of 30. In this context, it is essential to develop new cognitive tools integrating digital technologies and innovative approaches, which are indispensable for accurate diagnosis and monitoring of cognitive disorders in trisomy 21 patients. It was with this in mind that the ENDI (Evaluation Neuropsychologique dans la Déficience Intellectuelle) battery was designed. This neuropsychological battery comprises 15 subtests designed to assess language, memory, attention and executive skills. By analyzing changes in trisomy 21 patients performance over time, the neuropsychologist can detect early signs of AD. A pre-test of the ENDI battery is planned to evaluate subtest design, ergonomics and comprehension of instructions, and to identify any malfunctions. The observations gathered will enable the principal investigator to refine the digital design of the battery in collaboration with the publishing company.

ELIGIBILITY:
Inclusion Criteria:

Preliminary phase:

1. The inclusion criteria for the group of people with intellectual disabilities are as follows:

   * Participant who has received full information on the organization of the research and has not objected to his or her participation and to the use of his or her data.
   * Legal guardian of the participant, if applicable, who has received full information on the organization of the research and has not objected to participation and use of his/her data.
   * Age at inclusion: ≥ 25 and ≤ 65 years
   * Notion of intellectual disability in medical records
   * Access to the oral language of the participant with an intellectual disability: the subject's speech must be comprehensible to the evaluator and the subject must be able to understand simple statements. It is not possible to use an oral comprehension test (e.g. Token test by Renzi & Vignolo, 1962), as the norms achieved in healthy subjects would exclude almost all patients with intellectual disabilities, who have more limited language skills.
   * Enrolled in or benefiting from a social security scheme.
2. The inclusion criteria for the normotypic group are as follows:

   * Participant having received full information on the organization of the research and not having objected to his or her participation and to the use of his or her data.
   * Age at inclusion: ≥ 25 and ≤ 65 years
   * Affiliation with a social security scheme or beneficiary of such a scheme

Main phase:

Inclusion criteria are as follows:

* Participant with T21 who has received full information on the organization of the research and has not objected to participation and use of his/her data
* Legal guardian of the participant with T21, where applicable, who has received full information on the organization of the research and has not objected to his or her participation and the use of his or her data.
* Person with trisomy 21
* Age at inclusion: ≥ 25 and ≤ 65 years
* Access to the oral language of the participant with T21: the subject's speech must be comprehensible to the evaluator and the subject must be able to understand simple statements. It is not possible to use an oral comprehension test (e.g. Token test by Renzi & Vignolo, 1962), as the norms achieved in healthy subjects would exclude almost all patients with intellectual disabilities, who have more limited language skills.
* Membership of a social security scheme or beneficiary of such a scheme

Exclusion Criteria for both phases of the study are as follows:

* Disabling motor and/or sensory impairments preventing completion of the tests
* Insufficient command of the French language to complete the tests
* Severe general medical condition or alcoholism (habitual consumption of 3 drinks/day or history of alcohol withdrawal)
* History of stroke, severe head trauma, or cancer
* Change in long-term medication within 8 weeks prior to evaluation
* Refusal to participate by the subject and/or legal representative
* Individuals referred to in Articles L.1121-5 to L.1121-7 of the French Public Health Code:

  * Pregnant women, women in labor, or breastfeeding mothers
  * Individuals deprived of liberty by judicial or administrative decision
  * Individuals undergoing psychiatric treatment under Article L.3213-1 of the French Public Health Code

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normotypical volunteers, patients with intellectual disability, and Trisomie 21 patients (T21) will be recruited by psychologists during a consultation in the Geriatrics Department of the University Hospital of Nancy, either through the Memory Resource and Research Center outpatient clinic or the day hospital. Volunteers and patients are generally referred by their general practitioner or another hospital department.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Acceptability of individual subtests and the complete test battery | Through the study (completion of the full test battery), an average of 45 min
  Acceptability will be estimated by The average completion time for the complete ENDI battery
Acceptability of individual subtests and the complete test battery | Through the study (completion of the full test battery), an average of 45 min
  Acceptability will be estimated by the Average completion time for each subtest of the ENDI battery
Acceptability of individual subtests and the complete test battery | Through the study (completion of the full test battery), an average of 45 min
  Acceptability will be estimated by the Percentage of complete completion of each ENDI subtest
Acceptability of individual subtests and the complete test battery | Through the study (completion of the full test battery), an average of 45 min
  Acceptability will be estimated by the Percentage of subjects having completed all ENDI battery subtests

SECONDARY OUTCOMES:
The convergent validity of ENDI tests | Through the study, an average of 16 months
  Correlation coefficient between ENDI scores and scores on DSQIID-F questionnaire. Scoring scale for the DSQIID-F questionnaire is from 0 to 53
The convergent validity of ENDI tests | Through the study, an average of 16 months
  Correlation coefficient between ENDI scores and scores on BPSD-DS questionnaire . The Scoring scale for BPSD-DS questionnaire is : for each dimension, frequency is rated from 0 to 4 and severity from 0 to 3 .
The convergent validity of ENDI tests | Through the study, an average of 16 months
  Correlation coefficient between ENDI scores and score on ISDC questionnaire. Scoring scales for ISDC questionnaire is for each dimension, frequency is scored from 0 to 4, severity from 0 to 3 and impact from 0 to 5
The convergent validity of ENDI tests | Through the study, an average of 16 months
  Correlation coefficient between ENDI scores and scores of CAMCOG II questionnaire.
  The Scoring scale for CAMCOG II questionnaire is from 0 to 106, the lower the score, the greater the impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Nancy, Vandœuvre-lès-Nancy, Grand Est, France

REFERENCES:
- [Background] Hithersay R, Startin CM, Hamburg S, Mok KY, Hardy J, Fisher EMC, Tybulewicz VLJ, Nizetic D, Strydom A. Association of Dementia With Mortality Among Adults With Down Syndrome Older Than 35 Years. JAMA Neurol. 2019 Feb 1;76(2):152-160. doi: 10.1001/jamaneurol.2018.3616. PMID 30452522
- [Background] Coquelet A, Besozzi A, Roussel M, Lemetayer F. Evaluation neuropsychologique des adultes porteurs d'une trisomie 21 en Consultation memoire : quels outils ? Une revue de la litterature. Geriatr Psychol Neuropsychiatr Vieil. 2022 Mar 1;20(1):79-95. doi: 10.1684/pnv.2022.1025. French. PMID 35652846
- [Background] Coppus AW, Fekkes D, Verhoeven WM, Tuinier S, Egger JI, van Duijn CM. Plasma amino acids and neopterin in healthy persons with Down's syndrome. J Neural Transm (Vienna). 2007;114(8):1041-5. doi: 10.1007/s00702-007-0656-1. Epub 2007 Mar 31. PMID 17401539
- [Background] Carmeli E, Imam B, Bachar A, Merrick J. Inflammation and oxidative stress as biomarkers of premature aging in persons with intellectual disability. Res Dev Disabil. 2012 Mar-Apr;33(2):369-75. doi: 10.1016/j.ridd.2011.10.002. Epub 2011 Nov 25. PMID 22119683
- [Background] Burt DB, Aylward EH. Test battery for the diagnosis of dementia in individuals with intellectual disability. Working Group for the Establishment of Criteria for the Diagnosis of Dementia in Individuals with Intellectual Disability. J Intellect Disabil Res. 2000 Apr;44 ( Pt 2):175-80. doi: 10.1046/j.1365-2788.2000.00264.x. PMID 10898382
- [Background] Devenny DA, Zimmerli EJ, Kittler P, Krinsky-McHale SJ. Cued recall in early-stage dementia in adults with Down's syndrome. J Intellect Disabil Res. 2002 Sep;46(Pt 6):472-83. doi: 10.1046/j.1365-2788.2002.00417.x. PMID 12354318
- [Background] Startin CM, Hamburg S, Hithersay R, Al-Janabi T, Mok KY, Hardy J; LonDownS Consortium; Strydom A. Cognitive markers of preclinical and prodromal Alzheimer's disease in Down syndrome. Alzheimers Dement. 2019 Feb;15(2):245-257. doi: 10.1016/j.jalz.2018.08.009. Epub 2018 Nov 28. PMID 30503169
- [Background] Zis P, Strydom A. Clinical aspects and biomarkers of Alzheimer's disease in Down syndrome. Free Radic Biol Med. 2018 Jan;114:3-9. doi: 10.1016/j.freeradbiomed.2017.08.024. Epub 2017 Sep 1. PMID 28870521
- [Background] McCarron M, McCallion P, Reilly E, Dunne P, Carroll R, Mulryan N. A prospective 20-year longitudinal follow-up of dementia in persons with Down syndrome. J Intellect Disabil Res. 2017 Sep;61(9):843-852. doi: 10.1111/jir.12390. Epub 2017 Jun 29. PMID 28664561
- [Background] Lott IT, Head E. Down syndrome and Alzheimer's disease: a link between development and aging. Ment Retard Dev Disabil Res Rev. 2001;7(3):172-8. doi: 10.1002/mrdd.1025. PMID 11553933
- [Background] Lautarescu BA, Holland AJ, Zaman SH. The Early Presentation of Dementia in People with Down Syndrome: a Systematic Review of Longitudinal Studies. Neuropsychol Rev. 2017 Mar;27(1):31-45. doi: 10.1007/s11065-017-9341-9. Epub 2017 Mar 13. PMID 28289920
- [Background] Hartley D, Blumenthal T, Carrillo M, DiPaolo G, Esralew L, Gardiner K, Granholm AC, Iqbal K, Krams M, Lemere C, Lott I, Mobley W, Ness S, Nixon R, Potter H, Reeves R, Sabbagh M, Silverman W, Tycko B, Whitten M, Wisniewski T. Down syndrome and Alzheimer's disease: Common pathways, common goals. Alzheimers Dement. 2015 Jun;11(6):700-9. doi: 10.1016/j.jalz.2014.10.007. Epub 2014 Dec 12. PMID 25510383
- [Background] Godefroy O, Martinaud O, Verny M, Mosca C, Lenoir H, Bretault E, Roussel M. The dysexecutive syndrome of Alzheimer's disease: the GREFEX study. J Alzheimers Dis. 2014;42(4):1203-8. doi: 10.3233/JAD-140585. PMID 25024318
- [Background] Fortea J, Vilaplana E, Carmona-Iragui M, Benejam B, Videla L, Barroeta I, Fernandez S, Altuna M, Pegueroles J, Montal V, Valldeneu S, Gimenez S, Gonzalez-Ortiz S, Munoz L, Estelles T, Illan-Gala I, Belbin O, Camacho V, Wilson LR, Annus T, Osorio RS, Videla S, Lehmann S, Holland AJ, Alcolea D, Clarimon J, Zaman SH, Blesa R, Lleo A. Clinical and biomarker changes of Alzheimer's disease in adults with Down syndrome: a cross-sectional study. Lancet. 2020 Jun 27;395(10242):1988-1997. doi: 10.1016/S0140-6736(20)30689-9. PMID 32593336
- [Background] Rebillat AS, Hiance-Delahaye A, Falquero S, Radice G, Sacco S. The French translation of the dementia screening questionnaire for individuals with intellectual disabilities is a sensitive tool for screening for dementia in people with Down Syndrome. Res Dev Disabil. 2021 Nov;118:104068. doi: 10.1016/j.ridd.2021.104068. Epub 2021 Aug 28. PMID 34467872
- [Background] Dubois B, Touchon J, Portet F, Ousset PJ, Vellas B, Michel B. ["The 5 words": a simple and sensitive test for the diagnosis of Alzheimer's disease]. Presse Med. 2002 Nov 9;31(36):1696-9. French. PMID 12467149
- [Background] Grober E, Buschke H, Crystal H, Bang S, Dresner R. Screening for dementia by memory testing. Neurology. 1988 Jun;38(6):900-3. doi: 10.1212/wnl.38.6.900. PMID 3368071
- [Background] Krikorian R, Bartok J, Gay N. Tower of London procedure: a standard method and developmental data. J Clin Exp Neuropsychol. 1994 Dec;16(6):840-50. doi: 10.1080/01688639408402697. PMID 7890819
- [Background] DE RENZI E, VIGNOLO LA. The token test: A sensitive test to detect receptive disturbances in aphasics. Brain. 1962 Dec;85:665-78. doi: 10.1093/brain/85.4.665. No abstract available. PMID 14026018
- [Background] Rubenstein E, Hartley S, Bishop L. Epidemiology of Dementia and Alzheimer Disease in Individuals With Down Syndrome. JAMA Neurol. 2020 Feb 1;77(2):262-264. doi: 10.1001/jamaneurol.2019.3666. PMID 31657825
- [Background] Ball SL, Holland AJ, Treppner P, Watson PC, Huppert FA. Executive dysfunction and its association with personality and behaviour changes in the development of Alzheimer's disease in adults with Down syndrome and mild to moderate learning disabilities. Br J Clin Psychol. 2008 Mar;47(Pt 1):1-29. doi: 10.1348/014466507X230967. PMID 17681112